CLINICAL TRIAL: NCT02245841
Title: Efficacy and Safety of H.P. Acthar Gel for the Treatment of Refractory Cutaneous Manifestations of Dermatomyositis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Anthony Fernandez, MD, PhD, Md, PhD, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1015
Record Dates: First submitted 2014-09-11; First posted 2014-09-22 (Estimated); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Dermatomyositis; Juvenile Dermatomyositis
Keywords: dermatomyositis; Acthar gel
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.P Acthar Gel (Experimental): 80 U (1 mL) of H.P. Acthar gel via subcutaneous injection twice weekly for 24 weeks
  Interventions: Drug: H.P. Acthar Gel

INTERVENTIONS:
Drug: H.P. Acthar Gel — 80 U (1 mL) of H.P. Acthar gel via subcutaneous injection twice weekly for 24 weeks
  Other Names: Acthar Gel

SUMMARY:
This study will assess the safety and efficacy of H.P. Acthar gel for treating the cutaneous manifestations in patients with refractory classic dermatomyositis, juvenile dermatomyositis, and amyopathic dermatomyositis. Our hypothesis is that H.P. Acthar gel will be both safe and effective for such patients.

DETAILED DESCRIPTION:
Adult and juvenile dermatomyositis (DM) are systemic immune-mediated inflammatory diseases most commonly affecting the skin and musculoskeletal system. Amyopathic dermatomyositis is a subtype of dermatomyositis that affects only the skin and lacks the characteristic muscle involvement. Treatment of these conditions, in particular the cutaneous manifestations, is challenging and currently no universally effective single treatment exists. Many patients have cutaneous manifestations that are refractory to numerous medications.

H.P. Acthar gel (adrenocorticotropic hormone gel) received FDA approval for treatment of a variety of diseases, including dermatomyositis, in 1952. Despite this there is a paucity of clinical data concerning the efficacy of H.P. Acthar gel for treating dermatomyositis. Recently a small, retrospective case series describing significant improvement in both cutaneous and musculoskeletal symptoms in 5 patients with refractory dermatomyositis treated with H.P. Acthar gel was reported and has resulted in renewed interest in use of this medication in dermatomyositis patient (reference below). The proposed efficacy of H.P. Acthar gel has been attributed to its unique ability to induce production of endogenous cortisol, corticosterone, aldosterone, and to bind melanocortin receptors on lymphocytes and other cells to modulate immunologic responses.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older with refractory cutaneous symptoms related to either classic dermatomyositis (CD), juvenile dermatomyositis (JD), or amyopathic dermatomyositis(AD). Diagnosis will be based on either Bohan and Peter criteria (CD and JD) or Sontheimer's criteria (AD)
* Must have had a skin biopsy with histologic features consistent with dermatomyositis and current cutaneous manifestations consistent with dermatomyositis.
* Although not mandatory, patients with evidence of current or previous active myositis will be eligible for enrollment. Patients will be considered to have refractory disease if cutaneous manifestations exist despite treatment with steroids and at least one steroid-sparing systemic treatment commonly found to be useful in patients with dermatomyositis. These may include azathioprine, cyclosporine, mycophenolate mofetil, IVIG, methotrexate, cyclophosphamide, chlorambucil, sirolimus, adalimumab, infliximab and rituximab.
* Use of topical medications and sunscreen currently and in past will be noted but not weighed for assessment of refractory cutaneous disease.

Exclusion Criteria:

* Patients with dermatomyositis who have minimal-to-no active cutaneous features (focal involvement with less than 1% total body surface area involved or minimal modified CDASI activity score).
* Patients whose cutaneous findings are not consistent with dermatomyositis and/or have previous biopsy results suggestive of an alternative diagnosis
* Patients with inflammatory myositis other than dermatomyositis, such as polymyositis or inclusion body myositis.
* Patients with malignancy-associated dermatomyositis
* Patients with clear features of an overlap myositis
* Patients younger than 18 years old
* Patients with acutely active or chronic infections.
* Patients with uncontrolled diabetes, hypertension, cardiovascular, hepatic, or renal disease
* Pregnant or lactating females.
* Patients with any medical condition that is felt by the primary investigator to place the patient at unreasonable risk for adverse effects during treatment with H.P. Acthar.
* Hypersensitivity to H.P. Acthar, any of its components (allergy to pig-derived proteins)
* Patients with osteoporosis
* Patients who have had surgery within 8 weeks of screening
* Patients with a history of or current gastric ulcers
* Patients taking daily doses of systemic corticosteroids greater than the equivalent of 40mg prednisone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Fernandez, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited IPD will be shared within the publication.
Supporting Information: Study Protocol, SAP
Time Frame: CDSAI-A scores and adverse events at each study assessment point will be included and available in the publication indefinitely.
Access Criteria: Available to all.
URL: https://pubmed.ncbi.nlm.nih.gov/37941470/

REFERENCES:
- [Background] Levine T. Treating refractory dermatomyositis or polymyositis with adrenocorticotropic hormone gel: a retrospective case series. Drug Des Devel Ther. 2012;6:133-9. doi: 10.2147/DDDT.S33110. Epub 2012 Jun 11. PMID 22787386
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (first of two parts). N Engl J Med. 1975 Feb 13;292(7):344-7. doi: 10.1056/NEJM197502132920706. No abstract available. PMID 1090839
- [Background] Bohan A, Peter JB. Polymyositis and dermatomyositis (second of two parts). N Engl J Med. 1975 Feb 20;292(8):403-7. doi: 10.1056/NEJM197502202920807. No abstract available. PMID 1089199
- [Background] Gerami P, Schope JM, McDonald L, Walling HW, Sontheimer RD. A systematic review of adult-onset clinically amyopathic dermatomyositis (dermatomyositis sine myositis): a missing link within the spectrum of the idiopathic inflammatory myopathies. J Am Acad Dermatol. 2006 Apr;54(4):597-613. doi: 10.1016/j.jaad.2005.10.041. Epub 2006 Jan 23. PMID 16546580
- [Background] Euwer RL, Sontheimer RD. Amyopathic dermatomyositis: a review. J Invest Dermatol. 1993 Jan;100(1):124S-127S. doi: 10.1111/1523-1747.ep12356896. PMID 8423381
- [Background] Klein RQ, Bangert CA, Costner M, Connolly MK, Tanikawa A, Okawa J, Rose M, Fakharzadeh SS, Fiorentino D, Lee LA, Sontheimer RD, Taylor L, Troxel AB, Werth VP. Comparison of the reliability and validity of outcome instruments for cutaneous dermatomyositis. Br J Dermatol. 2008 Sep;159(4):887-94. doi: 10.1111/j.1365-2133.2008.08711.x. Epub 2008 Jul 4. PMID 18616782
- [Background] Yassaee M, Fiorentino D, Okawa J, Taylor L, Coley C, Troxel AB, Werth VP. Modification of the cutaneous dermatomyositis disease area and severity index, an outcome instrument. Br J Dermatol. 2010 Mar;162(3):669-73. doi: 10.1111/j.1365-2133.2009.09521.x. Epub 2009 Oct 26. PMID 19863510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | H.P Acthar Gel
Started | 19
Completed | 15
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 56 [35 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 19
Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI-A) [Median (Full Range); unit: units on a scale] — The CDASI-A score ranges from 0 to 100 with higher scores reflecting more severe disease activity.
  units on a scale | 19 [14 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cutaneous Dermatomyositis at 6 Months
Description: Change between baseline at 6 months in modified CDASI-A (Cutaneous Dermatomyositis Disease Area and Severity Index) scores at these timepoints.
  The CDASI-A score ranges from 0 to 100 with higher scores reflecting more severe disease activity.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 15
units on a scale | -9 [-18 to -5]
Statistical Analysis 1: Comparison: H.P Acthar Gel; Analysis performed was two-sided Wilcoxon signed rank test. Median differences with interquartile range are reported in outcome measure data; Test type: Superiority; p < .001, Wilcoxon signed rank test

2. Primary Outcome: Change in Physician's Global Assessment (PGA) Visual Acuity Score From Baseline to 6 Months
Description: Change from baseline to 6 months in Physician's Global Assessment (PGA) visual acuity score. Scores range from 0-10 with Higher scores reflecting severe disease activity.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 15
units on a scale | -1.9 [-2.5 to -1.2]
Statistical Analysis 1: Comparison: H.P Acthar Gel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon signed rank test

3. Secondary Outcome: Change From Baseline in Patient Assessment of Dermatomyositis at 6 Months.
Description: Change between baseline and 6 months in patient assessed "Global Skin Score" at these timepoints.
  The Global Skin Score ranges from 0 to 10 with lower 0 representing "worst sign condition imaginable" and 10 representing "perfect health".
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 15
units on a scale | 2 [.5 to 6]
Statistical Analysis 1: Comparison: H.P Acthar Gel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Wilcoxon signed rank test

4. Secondary Outcome: Change From Baseline in Patient Global Itch Score of Dermatomyositis at 6 Months
Description: Change between baseline and 6 months in patient assessed "Global Itch Score" at these timepoints.
  The Global Itch score ranges from 0 to 10 with higher scores reflect more severe itching.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 15
units on a scale | -1 [-5 to 1]
Statistical Analysis 1: Comparison: H.P Acthar Gel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.050, Wilcoxon signed rank test

5. Secondary Outcome: Change From Baseline in Patient Assessment of DLQI Dermatomyositis at 6 Months
Description: Change between baseline and 6 months in patient assessed Dermatology Life Quality Index (DLQI) scores at these timepoints.
  The DLQI ranges from 0 to 30 with higher scores implying more significant impact on quality of life.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | H.P Acthar Gel
Number analyzed (Participants) | 15
units on a scale | -5 [-11 to -4]
Statistical Analysis 1: Comparison: H.P Acthar Gel; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Wilcoxon signed rank test

6. Other Pre Specified Outcome: Number of Patients With Adverse Effects.
Description: Safety and tolerability of H.P. Acthar gel based on frequency and types of adverse effects.
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Patients With Change in Dose of Systemic Corticosteroids and/or Steroid-sparing Immunosuppressive Agents
Description: Median/mean change in dose of systemic corticosteroids and/or steroid-sparing immunosuppressive agents from initiation to completion of study
Time Frame: 6 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Number of Patients With Change in HbA1c
Description: Median/mean change in HbA1c
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 Months
Description: Standard definition
Arm/Group | H.P Acthar Gel
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 11/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | H.P Acthar Gel (N=19)
Difficulty Sleeping (General disorders) | 6
Weight Gain (General disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-07-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT02245841/Prot_SAP_000.pdf